CLINICAL TRIAL: NCT00311649
Title: Open Label Evaluation of H5N1 Vaccine at Vaccine Manufacturing Facilities
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05-0129; Influenza CVD 16000
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2007-03

CONDITIONS: Influenza
Keywords: H5N1, Influenza
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

INTERVENTIONS:
Biological: Inactivated Influenza A Vaccine A/H5N1

SUMMARY:
The purpose of this research is to study side effects and safety of a new H5N1 flu (bird flu) vaccine and to look at how well people's immune systems make antibodies to fight infection after they get the vaccine. Up to 300 healthy people who are working at Aventis Pasteur H5N1 virus vaccine production facility in Swiftwater, PA, during the flu season are being asked to participate. It is important for vaccine production workers to receive the vaccine in order to minimize the risk of this bird flu virus combining with the regular flu virus. Volunteers in this study will have a medical screening, 2 vaccinations a month apart, 2 blood sample collections (1 before and 1 after the vaccinations to compare), 5 clinic visits, and follow-up over 6 months. They will also complete a diary card and to write down their temperature once a day and any symptoms they have every day during the week after they get their second shot. They will also be asked to write down any drugs or medicines they take.

DETAILED DESCRIPTION:
The primary goal of this phase I/II, single center, open label study is to obtain additional safety and immunogenicity data on two 90 µg doses of H5N1. It is anticipated that this dose level will result in an acceptable proportion of subjects achieving a potentially protective postvaccination antibody titer combined with an acceptable safety profile. The purpose of the current study is to induce maximal anti-H5N1 titers as quickly as possible in order to protect at-risk personnel manufacturing a commercial-scale H5N1 vaccine under contract to the United States government. The study will be performed under the direction of investigators at the University of Maryland School of Medicine's Center for Vaccine Development. Volunteers will be enrolled, vaccinated, and followed at Sanofi Pasteur, in Swiftwater, PA. Up to 300 healthy vaccine production worker volunteers, aged 18 years and older, will receive 90 mcg of the influenza A/H5N1 vaccine by intramuscular injection. Volunteers will receive 2 doses of the vaccine separated by approximately 28 days. Serum HAI and neutralizing antibody titers will be assessed approximately 1 month after the second vaccine dose. Volunteers will be observed in the clinic for at least 15 minutes after each vaccination, and they will maintain a memory aid to record oral temperature and systemic and local adverse events (AEs) for seven days after each immunization. Volunteers will return to the clinic on Day 7 for AE and concomitant medication assessment, a targeted physical examination (if indicated), and review of the memory aid. Serum for immunogenicity evaluations will be obtained prior to the first vaccination (Day 0) and on Day 56. Primary study objectives are to: (1) determine the safety of subvirion inactivated A/H5N1 vaccine in healthy vaccine production workers adults; and (2) determine the immunogenicity of subvirion inactivated H5N1 vaccine in healthy adults approximately 1 month following receipt of two 90 mcg doses of vaccine. Primary study endpoints are: (1) adverse event (AE) or serious adverse event information (solicited in-clinic and via memory aids, concomitant medications, and periodic targeted physical assessment); (2) geometric mean titer (GMT) and frequency of 4-fold or greater increases in neutralizing antibody titers at two months after receipt of the first dose of vaccine; (3) GMT and frequency of 4-fold or greater increases in serum hemagglutination inhibition (HAI) antibody titers at 2 months after receipt of the first dose of vaccine; and (4) proportion of subjects achieving a serum neutralizing antibody titer of 1:40 against the influenza A/H5N1 virus 28 days after receipt of the second dose of vaccine (approximately Day 56).

ELIGIBILITY:
Inclusion Criteria:

1. Working in the production of H5N1 vaccine at Aventis Pasteur facilities at Swiftwater, Pennsylvania.
2. Male or nonpregnant female (as indicated by a negative urine pregnancy test prior to each dose of vaccine), aged 18 years and older.
3. Women of childbearing potential who are at risk of becoming pregnant must agree to practice adequate contraception (ie, barrier method, abstinence, and licensed hormonal methods) for the entire study period.
4. Is in good health, as determined by vital signs (pulse, blood pressure, oral temperature), medical history, and a targeted physical examination based on medical history.
5. Able to understand and comply with planned study procedures.
6. Provides informed consent prior to any study procedures and is available for all study visits.

Exclusion Criteria:

1. Has a known allergy to eggs or other components of the vaccine.
2. Has a known allergy or sensitivity to latex (in the stopper).
3. Is breastfeeding.
4. Is undergoing immunosuppression as a result of an underlying illness or treatment.
5. Has an active neoplastic disease or a history of any hematologic malignancy.
6. Is using oral or parenteral steroids, high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs.
7. Has a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
8. Has an acute illness, including an oral temperature greater than 100.4 degrees F, within 1 week of vaccination.
9. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to enrollment in this study, or expects to receive an experimental agent during the 6-month study period.
10. Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2005-11; Primary Completion 2006-09 (Actual); Study Completion 2006-09

CONTACTS AND LOCATIONS:
Locations (1):
- Sanofi Pasteur, Swiftwater, Pennsylvania, United States